CLINICAL TRIAL: NCT06428279
Title: Sexual Health in Cancer Patients: a Survey and Pilot Study of Psychosexual Therapy as a Non-pharmacological Supportive Care
Brief Title: Survey of Sexual Health in Cancer Patients
Acronym: S&C
Status: Completed | Type: Observational
Sponsor: Institut Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: IR-2024-001; 2024-A00387-40 (Other: ANSM)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Integrative Oncology
Keywords: Sexual health; Quality of life; Integrative oncology
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — survey

SUMMARY:
Sexual health, a vital aspect of the overall human health and a critical component of quality of life, can be negatively affected by cancer and cancer treatments. Although prevalence rates of sexual difficulties vary depending on several factors including primary diagnosis, treatment modality and methods of assessment, estimates rates are reported to range from 40% to 100%. Despite the abundant literature on sexuality and intimacy, communication about sexual health is often absent or inadequate between patients and health care providers. In this context, more research is needed to understand patients' priorities and needs for information about sexuality.

The purpose of this study is to assess the main difficulties faced by patients in their sexual life and to evaluate patient's satisfaction after having followed sessions of psychosexual therapy proposed at Rafaël Institute, France. The survey will be conducted using questionnaires developed specifically for this study. All questions will be coded through a Likert scale from 1 (strongly disagree) to 7 (strongly agree). Responses to each question will be analyzed with higher mean scores (>4) indicating main difficulties faced by patients in their sexual life. Patients will also express their positive or negative state of agreement regarding questions evaluating their satisfaction after following a program of psychosexual therapy. Approximately 200 patients will be invite to participated in this survey after provided oral consent.

DETAILED DESCRIPTION:
Sexual health, a vital aspect of the overall human health can be negatively affected by cancer and cancer treatments. Sexual dysfunctions affect the quality of life of an individual since sexual health is a critical component of overall quality of life. The World Health Organization (WHO) defines sexual health as "a state of physical, emotional, mental and social well-being in relation to sexuality; and not merely the absence of disease, dysfunction or infirmity". Indeed, regular sexual activity reduces stress, regularizes sleep cycle, and regulates our mental wellbeing as a whole.

Although prevalence rates of sexual difficulties vary among cancer patients and depend on several factors including primary diagnosis, treatment modality and methods of assessment, estimates rates can range from 40% to 100%. For example, in a French national survey focusing on sexual health of patients with colorectal or breast cancer two years after diagnosis, 54% of patients (235 of 435) reported to have a decrease in sexual desire and 61% had a decrease in frequency of intercourse.

Despite these problems have been well documented in the literature and in practice guidelines, many cancer survivors have limited access to high quality information on sexual health. Indeed, communication about sexual health is often absent or inadequate between patients and the medical team. Among barriers reported by health care providers for avoiding discussing this topic are lack of time, insufficient training, absence of awareness about the subject and unavailable access to integrative medicine solutions where they could send their patients. Cultural values, religious beliefs and social norms may also have significant implications.

Recognizing patients' sexual problems can help health care providers to offer appropriate integrative non-pharmacological interventions to different group of patients. In this context, more research is needed to understand patients' priorities and needs for information about sexuality. The purpose of this study is to assess the main difficulties faced by patients in their sexual life and to evaluate patient's satisfaction after having followed sessions of psychosexual therapy proposed at Rafaël Institute, France.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients
* adults aged > 18 years old

Exclusion Criteria:

* <18years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be adults aged 18 years old or older diagnosed with cancer and undergoing non-pharmacological supportive care during or after their standards cancer treatments at Rafael Institute
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
patients' satisfaction with their sexual lives | 1 month
  questionnaire

SECONDARY OUTCOMES:
identification of the main physiological and psychological difficulties encountered by patients in their sexual lives | 1 month
  questionnaire
patients perceived emotions | 1 month
  questionnaire
description of the impact of sex therapy sessions on the sexual health of the participants | 1 month
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Rafaël, Levallois-Perret, Institut Rafael, France

IPD SHARING:
Plan to Share IPD: Undecided